CLINICAL TRIAL: NCT02792270
Title: Effects Of Caloric Restriction On Post-Operative Complications In Sarcoma Patients Treated With Pre-Operative Radiation Therapy
Brief Title: Caloric Restriction In Sarcoma Patients Treated With Pre-Operative RT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Santiago Lozano-Calderon, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-485
Record Dates: First submitted 2016-05-16; First posted 2016-06-07 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Tumor Surgery
Keywords: Surgery
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caloric Restriction Diet (Experimental): Patients will meet with the Registered Dietitian to discuss calorie, protein, and fluid needs.The dietitian will calculate calorie needs.
  * Calorie needs will be reduced by 30%.
  * Protein needs will be estimated based on 0.8g/kg BW and then reduced by 70%.
  * Dietitian will educate participants on electrolytes and fluid intake based on the reduced food intake.
  Interventions: Other: Caloric Restriction Diet
- Normal Diet (No Intervention): Participant will follow a normal diet.

INTERVENTIONS:
Other: Caloric Restriction Diet — Two nutritional supplements, one from Ensure (Abbott Laboratories, Chicago, IL) and one from Boost (Nestle, Vevey, Switzerland) will be used for 3 days before surgery.
  The supplements are the Ensure Pre-Surgery Clear Carbohydrate Drink and the Ensure Original Nutrition Powder. The Original Nutrition Powder will be mixed with 8oz of water, oat milk, or almond milk. The proposed macronutrient profile for the 3 days of caloric restriction (CR) is less than 8% of calories from protein.
  Arms: Caloric Restriction Diet

SUMMARY:
This study is being conducted to decrease the rate of surgical wound complications. The investigators are studying the effects that caloric restriction has on decreasing the rate of surgical wound complications.

DETAILED DESCRIPTION:
The goal is to decrease the chance of having wound complications after surgery. Caloric Restriction has been found to be a natural modifier of surgical outcomes. Participants will be randomize into the arms Caloric Restriction Diet or Normal Diet.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Biopsy proven soft tissue sarcoma located in the lower extremities
* Patient to be treated with radiation therapy for a primary lower extremity soft tissue sarcoma or recurrent tumor after surgery, followed by surgical resection
* Karnofsky Score ≥ 60%
* Body Mass Index (BMI) ≥ 20 kg/m2
* Protein levels within normal limits within 45 days of enrollment
* Normal kidney and liver function within 45 days of enrollment
* Normal blood counts within 45 days of enrollment
* Normal chemistries within 45 days of enrollment

Exclusion Criteria:

* Current pregnancy and breast feeding
* Other cancers diagnosed within the last 5 years (in situ and/or invasive)
* Diabetes mellitus
* Current metformin therapy
* Other conditions may exclude participants from the study (e.g. intractable nausea/emesis, allergic reaction to shake, patient decides not to have surgery, any medical condition that prevents patient from having surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-06; Primary Completion 2026-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change In The Rate Of Physical Function By MSTS | Baseline, 6 weeks, 3 months and 6 months visits after surgery
  The Musculoskeletal Tumor Society Rating Scale (MSTS) is a clinician-based scoring system that is scored out of 35 points. A higher score indicates better physical function.
Change In The Rate Of Physical Function By TESS | Baseline, 6 weeks, 3 months and 6 months visits after surgery
  The Toronto Extremity Salvage Score (TESS) is a patient-reported scoring system that is scored out of 100 points. A higher score indicates better physical function.

SECONDARY OUTCOMES:
The Rate Of Wound Healing | 2 years
The Rate Of Wound Complications In The Protein Caloric Restriction (PCR) Versus Control Group | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Santiago A Lozano-Calderón, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No